CLINICAL TRIAL: NCT01864694
Title: Improving Dietary Behavior Through Tailored Messages
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Medical Center (Other)
Collaborators: University of Rhode Island (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 5R01HL081380 (NIH)
Record Dates: First submitted 2013-05-02; First posted 2013-05-30 (Estimated); Last update posted 2013-05-30 (Estimated); Status verified 2013-05

CONDITIONS: Cardiovascular Disease
Keywords: behavioral research; diet; health information systems
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- TLC-Diet (Experimental): Participants receive diet intervention through automated telephone system: TLC-Diet
  Interventions: Behavioral: TLC-Diet
- WEB-Diet (Experimental): Participants receive diet intervention through web-based system: WEB-Diet
  Interventions: Behavioral: WEB-Diet
- Control (Experimental): Assessment-only control group
  Interventions: Other: Assessment-only control

INTERVENTIONS:
Behavioral: TLC-Diet — Participants receive diet intervention through an automated telephone system
  Arms: TLC-Diet
Behavioral: WEB-Diet — Participants receive diet intervention through a web-based system
  Arms: WEB-Diet
Other: Assessment-only control — Assessment-only control
  Arms: Control

SUMMARY:
The aim of this study is to compare a Web-based system and a computer telephone system to determine their effectiveness in improving diet behaviors compared to each other and a control group.

DETAILED DESCRIPTION:
The aim of this study is to compare a Web-based system (WEB-DIET) and a computer telephone system (TLC [Telephone Linked Communications]-DIET) for affecting dietary behavior change. These interventions will target the same dietary behaviors (consumption of fat and fruits and vegetables). The behavior change strategies and content will be derived from the same behavior change theory (the Transtheoretical Model [TTM]). A representative sample of ~1200 adults from a large urban area will be recruited through a list-assisted telephone list which will be bought by the University of Rhode Island so that subjects can be randomized into one of three groups: a Web-based system (WEB- DIET), a computer telephone system (TLC [Telephone Linked Communications]-DIET), or assessment only control. The study hypotheses, which will be evaluated both at the end of the 6-month intervention period and at the end of 18-month follow-up (post-baseline) observation period, are: 1. TLC-DIET> Control 2. WEB-DIET> Control 3. WEB-DIET> TLC-DIET.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Be at risk with regard to saturated fat
* Have access to basic computer hardware and software
* Use the Internet regularly (defined as 1 times per week) and with basic proficiency
* Read and speak English at a fifth grade level
* Have access to a telephone and be able to use it independently.

Exclusion Criteria:

* Prescribed a diet that would conflict with a low saturated fat (e.g., a colectomy diet)
* Have a serious medical, psychiatric, or cognitive disease that would interfere with participation (e.g., cancer undergoing chemotherapy, psychotic disorder, Alzheimer's disease, etc.)
* If the individual does not use the Internet at least once a week

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1224 (Actual)
Dates: Start 2008-11; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Change in diet from baseline to 6 months, 6 months to 18 months, and baseline to 18 months | Baseline, 6 months, and 18 months
  Self-reported diet questionnaire to measure fat and fruits/vegetables

SECONDARY OUTCOMES:
Change in psychosocial variables from baseline to 6 months, 6 months to 18 months, and baseline to 18 months | Baseline, 6 months, and 18 months
  Additional theoretical variables, such as Stages of change, as measured by self-reported questionnaire
Change in diet variables from baseline to 6 months, 6 months to 18 months, and baseline to 18 months | Baseline, 6 months, and 18 months
  Additional diet variables, such as total calories, trans fat, and carotenoids, as measured by self-reported food frequency questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Robert H Friedman, MD, Principal Investigator — Boston University
Locations (1):
- Boston Medical Center, Boston, Massachusetts, United States